CLINICAL TRIAL: NCT01324401
Title: Oral Peanut Immunotherapy
Acronym: PNOIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Principal Investigator, Center for Immunology and Inflammatory Diseases; Director, Food Allergy Center, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010P000609
Record Dates: First submitted 2010-08-12; First posted 2011-03-29 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Peanut Allergy
Keywords: Peanut Allergy; Peanut Hypersensitivity
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The observational control arm (parallel for the first year) was then offered to cross over to active treatment
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The subjects randomized to the observational control group will have follow-up visits every 6 months. Each visit will involve a medical history and physical examination. These subjects are then offered to cross-over to active treatment.
- Peanut OIT (Experimental): The subjects randomized to the active treatment group will receive defatted peanut flour per protocol.
  Interventions: Drug: Peanut flour OIT

INTERVENTIONS:
Drug: Peanut flour OIT — Patients will receive daily escalating dosages (Peanut flour OIT) as determined in the modified rush phase as stated in the protocol. The dosage will be escalated until a daily dose of 4000 mg is reached. A Double-blind, placebo-controlled food challenge will then consist of two challenges performed on the same day. One challenge will consist of 7 doses of peanut given every 10-20 minutes in increasing amounts up to a total of 10 grams of whole peanut (5 grams of peanut protein) masked by inclusion in vehicle food. The other challenge will consist of placebo material given similarly.
  Arms: Peanut OIT

SUMMARY:
Peanut allergy is one of the most serious food allergies because of its life long persistence, and the potential for severe allergic reactions. Effective oral immunotherapy would benefit patients by reducing the likelihood that they will have life-threatening accidental allergic reactions. This research study is being done to develop an effective oral immunotherapy treatment for patients with peanut allergy.

DETAILED DESCRIPTION:
Our hypothesis is that chronic antigen exposure during peanut oral immunotherapy (OIT) will induce beneficial changes in the specific immune response, including: 1) anergy of IgE effector immune cells (e.g., mast cells, basophils) resulting in clinical desensitization; 2) induction of de novo, long lived (memory) B cell responses that antagonize specific IgE and confer immune tolerance. The investigators will test this hypothesis in the following specific aims:

1. Induce desensitization in peanut allergic subjects with peanut OIT and evaluate the safety of the peanut OIT desensitization protocol.
2. Induce long-standing tolerance in peanut allergic subjects with maintenance peanut OIT and evaluate the efficacy of allergen-specific testing to predict tolerance.
3. Longitudinally evaluate basophil and mast cell reactivity in subjects receiving peanut OIT and their relationship to the induction of desensitization.
4. Longitudinally evaluate the allergen-specific B-cell repertoire in subjects receiving peanut OIT and its relationship to the induction of tolerance.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of peanut allergy by a positive prick skin test to peanut (> 8 mm reaction wheal) or CAP FEIA >10 and a history of objective clinical symptoms within one hour after ingestion of peanuts
2. Ability to provide informed consent.
3. Males and females of all ethnic/racial groups between 7 and 21 years who are otherwise healthy.

Exclusion criteria:

1. Clinical history of a severe anaphylactic reaction known or suspected to be caused by ingestion of peanut that required treatment with 2 or more administrations of epinephrine or hospitalization
2. Moderate to Severe Asthma as defined using the Impairment or Risk Criteria of the current NHBLI Guidelines for the Diagnosis and Management of Asthma (http://www.nhlbi.nih.gov/guidelines/asthma/)
3. Poorly controlled Asthma as defined using the Control Criteria of the current NHBLI Guidelines for the Diagnosis and Management of Asthma (http://www.nhlbi.nih.gov/guidelines/asthma/)
4. Diagnosis of other severe or complicating medical problems
5. Autoimmune or chronic immune or gastrointestinal inflammatory conditions, including Celiac Disease, Inflammatory Bowel Disease and Eosinophilic Gastrointestinal Disorders
6. Primary Immune Deficiency
7. Use of beta blockers, angiotension converting enzyme inhibitors, or monoamine oxidase inhibitors
8. Women of childbearing potential who are pregnant, planning to become pregnant, or breastfeeding
9. Use within the past year of other systemic immunomodulatory treatment, including allergen immunotherapy, use of biologics with an immune target, including Xolair

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne G Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Food Allergy Center; Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control - Crossover: The subjects enrolled in the observational control group will have follow-up visits every 6 months. Each visit will involve a medical history and physical examination. After year 1, they will be offered to cross-over to active therapy.
- Peanut OIT: Peanut flour OIT: Patients will receive daily escalating dosages as determined in the modified rush phase as stated in the protocol. The dosage will be escalated until a daily dose of 4000 mg is reached. A Double-blind, placebo-controlled food challenge will then consist of two challenges performed on the same day. One challenge will consist of 7 doses of peanut given every 10-20 minutes in increasing amounts up to a total of 10 grams of whole peanut (5 grams of peanut protein) masked by inclusion in vehicle food. The other challenge will consist of placebo material given similarly.
Period: Overall Study
Arm/Group | Control - Crossover | Peanut OIT
Started | 4 | 26 (3 excluded from ITT analysis: 1 screen fail, 2 voluntary withdrawal pre-treatment)
Completed | 3 (one (1) could not tolerate minimum starting dose) | 20 (three (3) unable to complete due to adverse events)
Not Completed | 1 | 6
Not completed — Withdrawn before any treatment | 0 | 3
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Control - Crossover: The subjects enrolled in the observational control group will have follow-up visits every 6 months. Each visit will involve a medical history and physical examination. After year 1, they will have the opportunity to cross over to active therapy.
- Total: Total of all reporting groups
Arm/Group | Control - Crossover | Peanut OIT | Total
Number analyzed (Participants) | 4 | 26 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 26 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 12
  Male | 3 | 15 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 23 | 26
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 26 | 30

OUTCOME MEASURES:

1. Primary Outcome: Tolerance or Sustained Unresponsiveness
Description: The consumption of 5 grams of peanut protein during a double-blind placebo controlled food challenge without objective symptoms after one month of post treatment avoidance
Time Frame: at least 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Crossover | Peanut OIT
Number analyzed (Participants) | 4 | 23
Participants | 2 | 7

2. Secondary Outcome: Desensitization
Description: The consumption of 5 grams of peanut protein during an open food challenge without objective symptoms immediately post treatment
Time Frame: at least 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Crossover | Peanut OIT
Number analyzed (Participants) | 4 | 23
Participants | 3 | 19

ADVERSE EVENTS:
Time Frame: From Oct 2011 to July 2014
Arm/Group | Control - Crossover | Peanut OIT
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/23
Other Adverse Events (participants affected / at risk) | 4/4 | 23/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control - Crossover (N=4) | Peanut OIT (N=23)
Allergy: Skin/Oral pruritis (Immune system disorders) | 4 (68) | 18 (118)
Allergy: Multiple Symptoms (Immune system disorders) | 4 (18) | 22 (215)
GI: Abdominal Pain (Gastrointestinal disorders) | 4 (39) | 21 (191)
Resp: Wheeze/SOB (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 10 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No